CLINICAL TRIAL: NCT06913387
Title: Comparative Efficacy of Lipid Based Artificial Tears vs Aqueous Based Artificial Tears in Managing EDE: A 6 Week RCT
Brief Title: Comparative Efficacy of Lipid Based Artificial Tears vs Aqueous Based Artificial Tears in Managing EDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall23/792
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Evaporative Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipid Based Artificial Tears (Experimental)
  Interventions: Combination Product: Lipid Based Artificial Tears
- Aqueous Based Artificial Tears (Experimental)
  Interventions: Combination Product: Aqueous Based Artificial Tears

INTERVENTIONS:
Combination Product: Lipid Based Artificial Tears — 30 participants received lipid-based artificial tears (Recuro) in this study arm. The intervention involved the administration of RECURO EYE DROPS, which contain Sodium carboxymethylcellulose 0.5%. Participants were instructed to instill 1-2 drops in each eye, three times daily (morning, afternoon, and evening) throughout the 6-week trial period.
  Arms: Lipid Based Artificial Tears
Combination Product: Aqueous Based Artificial Tears — 30 participants received aqueous-based artificial tears (Softeal) in this study arm. The intervention involved the administration of SOFTEAL EYE DROPS, which contain Hydroxypropylmethyl Cellulose 0.3%. Participants were instructed to instill 1-2 drops in each eye, three times daily (morning, afternoon, and evening) throughout the 6-week trial period.
  Arms: Aqueous Based Artificial Tears

SUMMARY:
This research aimed to compare the effectiveness of a lipid-based artificial tear (Recuro) against an aqueous-based artificial tear (Softeal) in managing EDE symptoms and signs.

DETAILED DESCRIPTION:
This prospective, double-blind, randomized clinical trial was conducted at Mughal Eye Hospital, Lahore. A sample size of 60 participants (30 per group) was determined using G*Power. Participants (18-55 years, both genders) were assigned 1:1 to Recuro or Softeal for 6 weeks using block randomization (block size 4) generated by Research Randomizer. Primary outcomes included OSDI (Ocular Surface Disease Index) and SANDE (Symptom Assessment in Dry Eye) scores; secondary outcomes were Tear Break-Up Time (TBUT), Schirmer's test, and Meibomian gland expression.

ELIGIBILITY:
Inclusion Criteria:

* Adults (both genders) aged 18-55 years diagnosed with evaporative dry eye (EDE).
* Willingness to adhere to the prescribed treatment regimen (lipid-based or aqueous-based artificial tears).
* Include patients with a history of dry eye symptoms for at least 1-3 months.
* Ocular Surface Disease Index (OSDI) score ≥13, indicating the presence of mild to severe dry eye symptoms.
* Patients with tear break-up time (TBUT) <10 seconds, indicating tear film instability.

Exclusion Criteria:

* Use of any topical ophthalmic medications (e.g., lubricants, anti-inflammatory drugs, or cyclosporine) for dry eye within the last 1 month.
* Active ocular infection or inflammation (e.g., conjunctivitis, uveitis).
* History of ocular surgery or trauma within the past 6 months.
* Participants currently wearing contact lenses or those who have worn contact lenses in the past three months.
* Systemic conditions known to impact ocular surface health, such as uncontrolled diabetes, autoimmune disorders, or Sjögren's syndrome.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | 12 Months
  Assesses dry eye symptom frequency and impact on vision-related activities. Score ranges from 0-100.
  Scoring: 0-12 (Normal), 13-22 (Mild dry eye), 23-32 (Moderate dry eye), ≥ 33 (Severe dry eye).
SANDE Questionnaire (Symptom Assessment in Dry Eye) | 12 Months
  Measures the frequency and severity of dry eye symptoms. Score ranges from 0-100.
  Scoring: Higher scores indicate more severe and frequent symptoms
Meibum Test Score | 12 Months
  This score quantifies meibomian gland health and lipid secretion based on meibum quality and expressibility. It is derived from the assessment of 5 central glands in the lower eyelid.
  Scoring: Each assessed gland is scored from 0-3, resulting in a total Meibum Test Score for each eye ranging from 0-15.
  * Meibum Test Score Key (Per Gland):
  * 0: Clear meibum, no blockage (Healthy function)
  * 1: Cloudy meibum, mild dysfunction
  * 2: Thickened meibum, partial blockage
  * 3: No meibum expressed, severe obstruction
  * Interpretation: Lower total scores indicate healthier meibomian gland function and better meibum quality/expressibility.
Tear Break-up Time (TBUT): ( without anesthesia) | 12 months
  Measures tear film stability by observing the time (in seconds) until the first dry spot appears on the cornea after blinking.
  Scoring: TBUT <10 seconds is indicative of tear film instability and often associated with dry eye.
Schirmer Test I | 12 Months
  Measures tear volume by assessing the length of wetting on a filter paper strip (in millimeters) after 5 minutes, without anesthesia.
  Scoring: ≥10 mm (Normal Tear Production),
  * 5-9 mm: Mild to Moderate Tear Deficiency (or decreased production), often associated with mild to moderate dry eye
  * <5 mm: Severe Tear Deficiency (or significantly decreased production), indicative of severe dry eye

CONTACTS AND LOCATIONS:
Locations (1):
- Mughal eye Hospital Johar town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No